CLINICAL TRIAL: NCT00446602
Title: A Phase 2, Randomized, Open-Label Study To Assess The Safety And Efficacy Of Weekly (QW) Or Once Every Two Week (Q2W) Dosing Of Epoetin Alfa (PROCRIT) in Anemic Subjects With Low- or Intermediate-1 Risk Myelodysplastic Syndromes (MDS)
Brief Title: A Phase 2 Study to Evaluate the Safety and Effectiveness of Once Weekly or Once Every Two Week Dosing of Epoetin Alfa in Anemic Patients With Low- or Intermediate-1 Risk Myelodysplastic Syndromes (MDS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to company decision to focus resources on a larger, controlled study in this patient population.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013198
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2011-06

CONDITIONS: Myelodysplastic Syndromes; Anemia
Keywords: PROCRIT; Epoetin alfa; Myelodysplastic Syndromes; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 001 (Experimental): Epoetin alfa Type=exact unit=units number=80 000 form=solution for injection route=subcutaneous use once every week or once every 2 weeks.
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — Type=exact, unit=units, number=80,000, form=solution for injection, route=subcutaneous use, once every week or once every 2 weeks.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of PROCRIT (Epoetin alfa) 80,000 Units given once weekly or 80,000 Units given once every two weeks in anemic patients with Low- or Intermediate-1 risk Myelodysplastic Syndromes (MDS).

DETAILED DESCRIPTION:
This is a randomized (patients are assigned to a type of treatment by chance), open-label (both the patient and the physician know what treatment is being given), multi-center study in approximately 100 anemic patients with Low- or Intermediate-1 risk Myelodysplastic Syndromes (MDS). Patients with a diagnosis of MDS via bone marrow aspirate and biopsy according to World Health Organization (WHO) Criteria or French-American-British (FAB) Classification, and International Prognostic Scoring System (IPSS) of Low- or Intermediate-1 risk disease (<=10% bone marrow blasts), a baseline hemoglobin (Hb) < 10.0 g/dL [defined as the average of at least 2 measurements (not influenced by red blood cell (RBC) transfusions for at least 1 week) greater than or equal to 1 week apart], and who meet all other inclusion/exclusion criteria will be randomized to receive PROCRIT (Epoetin alfa) 80,000 Units under the skin (sc) once weekly (qw ) or 80,000 Units sc once every 2 weeks (q2w).

The total study duration is up to 30 weeks, including up to a 2-week screening phase, a 24-week dosing phase, a follow-up visit according to the patient's assigned visit schedule, and a 4-week safety follow-up phase.

Beginning at Week 13, and every week thereafter, patients will be assessed for Erythroid Response. Overall Erythroid Response (OER) (as per the 2000 International Working Group (IWG) Criteria) including Major and Minor Erythroid Responses is defined as: Major Erythroid Response: Having sustained one of the following criteria over a minimum of 8 weeks: >2 g/dL rise in hemoglobin (Hb), OR transfusion independence for patients who were RBC transfusion dependent (defined as requiring 4 or more red blood cell (RBC) units within 8 weeks prior to the first dose of PROCRIT (Epoetin alfa) ) at baseline. Minor Erythroid Response is defined as: Having sustained one of the following criteria over a minimum of 8 weeks: 1-2 g/dL rise in Hb, OR 50 to <100% transfusion reduction for patients who were RBC transfusion dependent (defined as requiring 4 or more RBC units within 8 weeks prior to the first dose of PROCRIT (Epoetin alfa)) at baseline.

Overall Erythroid Response (OER) (as per the 2006 Modified IWG Criteria) is one of the secondary endpoints of the study and is defined as: Having sustained one of the following criteria over a minimum of 8 weeks: >= 1.5 g/dL rise in Hb, OR Reduction in transfusion requirements by at least 4 RBC units for patients who were RBC transfusion dependent (defined as requiring 4 or more RBC units within 8 weeks prior to the first dose of PROCRIT (Epoetin alfa) at baseline. Only RBC transfusions given for a Hb of <= 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation.

Fatigue assessments [Brief Fatigue Inventory (BFI) and Medical Outcome Survey (MOS) Short Form-36 (SF-36)] will be completed by patients at baseline (Day 1/Week 1), Week 9, Week 13, and at end of study. In addition, a Global Rating of Change in Level of Fatigue (single-item question) will be completed by patients at Week 13 and end of study.

Safety evaluations will be performed at specified intervals during the study. Hb, hematocrit (Hct), and blood pressure will be monitored weekly. Clinical safety will be assessed by the incidence and severity of adverse events, clinical laboratory tests (Hb and Hct), vital signs and physical examinations during the study period.

Patients will be randomized in a 1:1 ratio to receive PROCRIT (Epoetin alfa) 80,000 Units given under the skin once a week or 80,000 Units given under the skin once every 2 weeks. Dose adjustments will be made (i.e., dose increased or decreased, frequency decreased, or doses withheld) in response to Hb monitoring throughout the study and in order to maintain a Hb level in the target range of 11 to 12 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Myelodysplastic Syndromes (MDS) via bone marrow aspirate and biopsy according to World Health Organization (WHO) Criteria or French-American-British (FAB) Classification. All WHO and FAB subtypes of MDS are potentially eligible, provided the subject's International Prognostic Scoring System (IPSS) score is Low- or Intermediate-1 [with the exception of chronic myelomonocytic leukemia (CMML)]
* Documentation of IPSS score of Low- or Intermediate-1 risk disease (<= 10% bone marrow blasts), based on bone marrow aspirate, biopsy, and cytogenetics, within 12 weeks prior to study entry
* Baseline hemoglobin (Hb) value of <10 g/dL [defined as the average of at least 2 measurements [(not influenced by red blood cell (RBC) transfusions for at least 1 week) >= 1 week apart]. The Hb level prior to the first dose of PROCRIT (Epoetin alfa) cannot be > 10.5 g/dL.

Exclusion Criteria:

* No anemia due to factors other than MDS (including hemolysis or gastrointestinal bleeding)
* No proliferative (White Blood Cells (WBC) >= 12,000/mm3) chronic myelomonocytic leukemia (CMML)
* No history of (within 12 months) deep venous thrombosis [(DVT), includes proximal and distal], pulmonary embolism (PE), or other venous thrombosis. Prior superficial thrombophlebitis is not an exclusion criterion
* No history of (within 6 months) cerebrovascular accident [(CVA), includes ischemic, embolic and hemorrhagic], transient ischemic attack (TIA), myocardial ischemia [includes Unstable Angina, Q wave Myocardial Infarction (QwMI) and non-Q wave Myocardial Infarction (NQMI)], or other arterial thrombosis
* No prior Erythropoietin Receptor Agonist (ERA) treatment within 4 weeks prior to the first study dose
* No prior ERA treatment failure (defined as having shown no Hb response or a Hb response <1 g/dL after at least 6 weeks of ERA treatment) with minimum dose of Epoetin alfa 40,000 Units/week or Darbepoetin alfa 150 mcg/ week.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of patients (POP) in each treatment group achieving an Overall Erythroid Response (OER) [as per the 2000 International Working Group (IWG) Criteria] by Week (Wk) 13 of the study.

SECONDARY OUTCOMES:
Proportion of patients (POP) w/OER by Wk 24 & study end; time and duration of OER; POP w/OER by Wk 13 & 24 (2006 IWG criteria);time to achieve Hb 11 g/dL; score change of BFI & SF-36 from baseline to study end;POP remaining RBC-transfusion free by Wk 24

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.